CLINICAL TRIAL: NCT03091998
Title: A Phase I Trial to Determine Safety and Efficacy of Chronic Subcu Administration of CD-NP in Heart Failure Patients With Left Ventricular Assist Device Support
Brief Title: Subcu Administration of CD-NP in Heart Failure Patients With Left Ventricular Assist Device Support
Acronym: CD-NP/LVAD
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No funding available
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Tomoko Ichiki, M.D., Ph.D., Associate Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB # 16-004850
Record Dates: First submitted 2017-03-09; First posted 2017-03-27 (Actual); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Heart Failure; Left Ventricular Assist Device; Natriuretic Peptide
MeSH Terms: conditions — Heart Failure | interventions — cenderitide; Saline Solution

STUDY DESIGN:
Intervention Model Description: Injection of CD-NP vs Placebo
Who Masked: Participant, Care Provider, Investigator
Masking Description: The Research Pharmacists will manage the randomization of the study and release information at the conclusion, once all participants have been recruited and completed study measures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Drug (CD-NP) (Active Comparator): Participants will receive a single subcutaneous injection of CD-NP (5 ug/kg) for 3 days running
  Interventions: Drug: CD-NP
- Placebo (saline) (Placebo Comparator): Participants will receive a single subcutaneous injection (~1 mL) of normal saline for 3 days running
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CD-NP — Participants will receive a subcutaneous injection of CD-NP (5 mcg / kg) daily for 3 days
  Other Names: Cenderitide
  Arms: Study Drug (CD-NP)
Other: Placebo — Participants will receive an ~ 1mL subcutaneous injection of normal saline, in lieu of Study Drug, for 3 days
  Other Names: 0.9% normal saline
  Arms: Placebo (saline)

SUMMARY:
The worldwide use of left ventricular assist devices (LVAD), which is mechanical device to improve hemodynamic function, has improved the outcomes of severe heart failure (HF) patients leading to the continued annual increase in the number of LVAD implantations. However LVAD support still results in major complications such as renal failure or gastrointestinal bleeding. The investigators hypothesize that such major complications may be due to endothelial dysfunction induced by the lack of pulsatility, which may be improved by an innovative designer natriuretic peptide, CD-NP. They have demonstrated its favorable actions in animal models as well as humans, and tested its safety in LVAD patients. They hypothesize that CD-NP will have renal and endothelial protective actions through its receptor GC-A and GC-B. Thus, the investigators will test their hypothesis with a highly translational approach to examine CD-NP's role in endothelial and renal protection.

The aim is to determine safety and tolerability together with cGMP activating, neurohumoral modulating and renovascular protective properties of chronic subcutaneous delivery of CD-NP compared to placebo in stable LVAD patients for 3 days.

DETAILED DESCRIPTION:
Stable patients with LVAD implantation (3 months s/p implantation) will undergo 3-day testing in the Mayo Clinic's Clinical Research and Trials Unit. They will undergo daily subcutaneous injection of CD-NP, or placebo, for 3 days with hemodynamic monitoring, ECHO, endothelial function assessment, and renal blood flow monitoring. Blood and urine samples will also be collected and assayed.

ELIGIBILITY:
Inclusion Criteria:

* Male and non-pregnant/post-menopausal/sterile females, ages 18-90, in end-stage HF with LVAD support who are stable in the healed stage at least 3 months from the LVAD implant (Destination therapy only) (the post-menopausal state is defined as the absence of menses for ≥ 1 year or serum follicle-stimulating hormone ≥ 20 IU/L; sterilization in the female is defined as bilateral tubal occlusion for ≥ 6 months, bilateral oophorectomy, or complete hysterectomy)
* Be willing to provide informed consent.
* All cardiac medications must be at stable doses 4 weeks prior to enrollment.

Exclusion Criteria:

* Known allergy or other adverse reactions to exogenous natriuretic peptides (CD-NP or its components, nesiritide, other natriuretic peptides, or related compounds).
* Women who are pregnant, or breast-feeding.
* Having received nesiritide within 7 days prior to entry into the study.
* Having received any investigational drug or device within 30 days prior to entry into the study.
* Clinically unstable patients (e.g. mean blood pressure < 70 mmHg, ongoing requirement for vasopressors, or mechanical ventilation).
* Recent hospitalization for decompensated HF or recent defibrillation for cardiac resuscitation within 30 days prior to randomization.
* Patients with guarded prognosis who are unlikely to derive meaningful benefit from CD-NP.
* Presence of cardiac lesions or comorbidities that may contraindicate the use of natriuretic peptides, such as clinically significant cardiac valvular stenosis, hypertrophic cardiomyopathy, restrictive cardiomyopathy, constrictive pericarditis, primary pulmonary hypertension, or uncorrected congenital heart disease that contraindicates the use of vasodilators.
* Symptomatic carotid artery disease, known critical carotid stenosis, or stroke within the past 3 months
* Requirement of pressors for maintenance of blood pressure.
* Intra-aortic blood pump use.
* Severe aortic or mitral stenosis or significant LV outflow tract obstruction.
* Clinically significant renal artery stenosis > 50%
* Baseline hemoglobin < 9.0 g/dl.
* Serum sodium < 130 mEq/L, potassium < 3.6 mEq/L, or magnesium < 1.5 mEq/L.
* Elevated aspartate aminotransferase (AST) or alanine aminotransferase (ALT) at least 5 times the upper limit of normal or bilirubin at least 5 times the upper limit of normal
* Creatinine clearance (CrCl) < 30 ml.min-1.1.73m-2, as calculated by Cockcroft-Gault formula(67) and adjusted for body surface area within 3 months or requirement for dialysis.
* Written history of alcohol or drug abuse within the past 6 months.
* Inability to communicate effectively with study personnel.
* BMI >40

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09-30 (Estimated); Primary Completion 2019-05-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Hypotension | 2 weeks
  To assess safety and tolerability (without symptomatic hypotension or mean blood pressure <70 mmHg) of chronic continuous subcutaneous infusion administration of CD-NP.

SECONDARY OUTCOMES:
Pharmacokinetic Outcome Characterization | 2 weeks
  Area under the plasma concentration versus time curve (AUC) assessed by plasma CD-NP and cGMP
Renal Function | 2 weeks
  Estimated GFR from creatinine clearance and
Endothelial function | 2 weeks
  Measurement by Reactive Hyperemia-peripheral arterial tonometry (RHI)

CONTACTS AND LOCATIONS:
Overall Officials: Tomoko Ichiki, M.D.Ph.D., Principal Investigator — Mayo Clinic

IPD SHARING:
Plan to Share IPD: No